CLINICAL TRIAL: NCT06003920
Title: Outcomes of a Small Process Group on Medical Students' Grit, Resilience, and Stress: A Quasi-experimental Pilot Study
Brief Title: Outcomes of a Small Process Group on Medical Students' Grit, Resilience, and Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University of Health Sciences (Other)
Responsible Party: Principal Investigator, Edie Sperling, Assistant Professor and Vice-Chair, Medical Anatomical Sciences, Western University of Health Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1902099
Record Dates: First submitted 2023-07-31; First posted 2023-08-22 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Stress
Keywords: medical students; stress; grit; resilience

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: Interventionist was blinded to which group participants were also research participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Process Group (Experimental): Medical students enrolled in the small process group, led by psychiatrist.
  Interventions: Behavioral: Process group
- Control Group (No Intervention): Medical students from the same cohorts, not enrolled in the small process group.

INTERVENTIONS:
Behavioral: Process group — The medical student process group served as a space for students to gain increased self-awareness through guided exploration of the psychodynamic processes.
  Arms: Process Group

SUMMARY:
The incidence of burnout and mental ill-health begins very early in medical school and continues to be high throughout training. Medical students are under high amounts of stress, which often becomes chronic, and can lead to both physical and psychological issues as a student, resident, and physician. Chronic stress and burnout in medical students are not a new phenomenon, but recent research has highlighted the worsening mental health of medical students, with as high as three-quarters of students reporting mental ill-health. It is vital that ways are found to reduce burnout and assist in improving the mental health of medical students. This quasi-experimental study aimed to assess the effect of a small process group vs. a control group of preclinical medical students on their stress, resilience, and grit.

DETAILED DESCRIPTION:
The investigators assessed the effects of a year-long small process group intervention, led by a psychiatrist, which aimed to improve self-awareness, mindfulness, and resilience in first and second-year medical students. Students self-selected into the process group, and the same number were randomly recruited as controls from the rest of the preclinical student body. The psychiatrist who led the groups was blinded to student participation in the study. Students in the process and control groups were surveyed with the Perceived Stress Scale, the Connor-Davidson Resilience Scale, and the Grit Scale in September 2022, and again after nine months and 25 sessions, in May 2023, after the academic year. Statistical analysis was done with R Studio. Bandura's theory of self-efficacy was used to conceptualize the study. Recruitment was done by email, as was data collection. The intervention included guided exploration of the psychodynamic process, group dynamic theory, cognitive behavioral therapy, dialectical behavioral therapy, boundaries, and empathy.

ELIGIBILITY:
Inclusion Criteria:

1. The participant must be an enrolled student at the College of Osteopathic Medicine of the Pacific-NW
2. Participant must be in their first or second year of medical school
3. Participant must be at least 18 years of age
4. Participant must self-select into either the intervention group or control group
5. Participant must sign informed consent

Exclusion Criteria:

1. Data will be excluded if a student goes on a LOA during the course of the year
2. Data will be excluded if a student does not attend a minimum of 12 out of 25 small group sessions
3. Student does not give informed consent
4. Student withdraws consent at any time

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-06-24 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Scale-14 | 34 weeks
  Stress measured on a 0-56 scale; higher number means more stress. Each of the 14 questions is measured on a 0-4 scale of 0 = Never, 1 = Almost Never, 2 = Sometimes, 3 = Fairly Often, 4 = Very Often.
Connor-Davidson Resilience Scale-25 | 34 weeks
  Resilience is measured on this 25-item scale, with higher numbers meaning more resilience. The score can range between 0 and 100. Each item has anchors from 0-4.
The Grit Scale | 34 weeks
  The original 12-item grit scale was used to measure grit; each items is rated 1-5, then scores are summed and divided by 12, so the final score is between 1-5. Higher scores mean more grit.

SECONDARY OUTCOMES:
Medication or diagnosis change | 34 weeks
  Change in anti-depression, anti-anxiety, or other mental health medications or diagnoses on a binary yes/no scale.

CONTACTS AND LOCATIONS:
Overall Officials: Edie L Sperling, DPT, Principal Investigator — Western University of Health Sciences
Locations (1):
- College of Osteopathic Medicine of the Pacific - Northwest, Lebanon, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
All anonymized demographic and outcome data will be shared in an open-access data repository.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Study protocol and SAP will be shared with results. Informed consent is shared here.
Access Criteria: Open access.
URL: https://www.kaggle.com/datasets/esperling/stress-grit-and-resilience-in-medical-students

DOCUMENTS (1):
  • Informed Consent Form (2022-06-24): https://cdn.clinicaltrials.gov/large-docs/20/NCT06003920/ICF_000.pdf